CLINICAL TRIAL: NCT01317355
Title: Prevalence of Multiple Symptoms in Cancer Patients a Cross Sectional Prospective Multi Center Study
Brief Title: Multiple Symptoms in Cancer Patients a Cross Sectional Multi Center Study
Acronym: ProKID
Status: Completed | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Patrick Jahn, Dr. rer. medic. Patrick Jahn, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: ProKID
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Cancer
Keywords: Cancer; Symptom burden; Symptom cluster; Distress; Pain; Fatigue; Sleep disorder; HRQoL
MeSH Terms: conditions — Neoplasms; Syndrome; Pain; Fatigue; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cancer patients: in and out patients of 5 German university hospitals currently undergoing cancer treatment

SUMMARY:
This study will assess the occurrence of multiple symptoms in cancer patients of 5 German university hospitals. Primary goal of the study is to assess the prevalence of multiple symptoms and related symptom clusters (e.g. pain, fatigue and sleep disorder).

DETAILED DESCRIPTION:
Oncology patients experience a variety of symptoms as a result of disease and/or treatment. They often report co-occurrence of symptoms and functional impairments (Miaskowski 2007). To evaluate the prevalence of symptoms and identify symptom clusters and the influence of multiple symptoms on HRQoL, in and out patients of 5 German university hospitals currently undergoing cancer treatment are recruited. These patients are asked to complete the following instruments: Distress thermometer, health related quality of life questionnaire (EORTC QLQ C30) and MD. Anderson Symptom Inventory (MDASI (German version). In a subgroup of two participating hospitals patients, that score ≥ 3/10 (MDASI-subscales for pain, fatigue and/or sleep disorder) are asked to complete additional questionnaires: Brief Pain Inventory (BPI), Multidimensional Fatigue Inventory (MFI), Pittsburgh Sleep Quality Index (PSQI). The information gained will not be accessible for doctors in charge of the treatment and therefore not influence or alter the participants' treatment regimes.

Primary endpoint of the study is to assess the prevalence of multiple symptoms and related symptom clusters (e.g. pain, fatigue and sleep disorder). Secondary endpoints are: symptom burden (intensity of symptoms and functional impairments), impact of symptom burden on HRQoL.

The investigators aim to approve the value of standardized assessment of symptoms in clinical cancer care settings as an important precondition of early treatment and supportive care.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients (ICD 10)
* 18 to 80 years of age
* ongoing treatment
* informed consent

Exclusion Criteria:

* not speaking and writing German

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: in and out cancer patients of 5 German university hospitals currently undergoing cancer treatment
Sampling Method: Probability Sample
Enrollment: 697 (Actual)
Dates: Start 2010-06; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Symptom burden (intensity & functional impairment) (MDASI) | 24 hours

SECONDARY OUTCOMES:
Distress thermometer | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Margarete Landenberger, Prof.Phd, Principal Investigator — Department for Health and Nursing Science, Medical Faculty, Martin-Luther-University Halle-Wittenberg
Locations (1):
- Department for Health and Nursing Science, Medical Faculty, Martin-Luther-University Halle-Wittenberg, Halle, Saxony-Anhalt, Germany